CLINICAL TRIAL: NCT04928924
Title: Functional Biomechanical Analysis in Immediate Post-Operative Period Following Total Hip Arthroplasty - A Pilot Study
Brief Title: Immediate Post-THA Functional Assessment
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Golden Jubilee National Hospital (Other Government)
Collaborators: Stryker GI Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-07
Record Dates: First submitted 2021-06-03; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Arthritis of Hip
Keywords: Total Hip Arthroplasty; Total Hip Replacement; biomechanical assessment; gait analysis; movement analysis
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — We will be observing patients who have undergone surgical replacement of arthritic hip with an implant.

SUMMARY:
The objective of this study is to investigate the feasibility of functional 3D biomechanical assessment and EMG analysis of gait and a sit to stand tasks in the immediate post-operative phase following total hip arthroplasty.

DETAILED DESCRIPTION:
Functional recovery is often an important priority for patients undergoing total hip arthroplasty (THA) and it is thought that abnormal biomechanics may be an obstacle to full recovery of physical function. While there has been extensive research on the biomechanics of gait and other activities of daily living following THA, the earliest reported post-operative assessment of function using 3D motion analysis for kinematics and kinetics has been at 6 weeks post-surgery. There is a paucity of data from the immediate post-operative phase prior to patient discharge from hospital.

In recent years there has been an increase in initiatives such as fast-track or enhanced post-operative recovery programs following joint arthroplasty, with the aim being an early return to function and shorter hospital length of stay whilst maintaining the low morbidity and mortality and high satisfaction rates typically associated with THA. There has also been continued research and developments on improving the THA procedure and while initial focus on improving THA surgery centred on implant design, materials and fixation to bone, there has been increased attention to surgical approach. In the last 10 years the use of minimally invasive surgical techniques has become more widespread due to the potential reported benefits. These include a shorter incision length, reduced muscle damage, reduced pain and less bleeding. When combined, these benefits may lead to reduced length of hospital stay and earlier return to function.

With so much focus centred on early return to function, there is a need to objectively measure function in the immediate post-operative phase. This would allow us to evaluate the effect of minimally invasive surgical approaches and enhanced recovery programs, which are primarily centred on early recovery from surgery. The use of 3D motion capture technology allows for accurate assessment of joint movement in three planes during dynamic movements and has been used extensively in the evaluation of function in patients with significant hip pathology before and after total hip arthroplasty. As aforementioned, to date the earliest post-operative motion analysis has been at 6 weeks after THA. Similarly, the earliest reported time point for muscle activation analysis using EMG is 6 weeks post THA. The aim of this study is assess the feasibility of 3D motion analysis including EMG in the immediate post-operative phase following THA in a hospital which incorporates an Enhanced Recovery After Surgery (ERAS) program as part of routine clinical care. This pilot project will guide development of future protocols which require early post-operative 3D biomechanical analysis.

For the purposes of this study the investigators define the immediate post-operative time point as the day the patient is discharged from the inpatient rehabilitation team and therefore deemed "safe" to mobilise independently by the ward physiotherapists.

Subject recruitment and retention will be closely monitored throughout the trial, allowing us to measure recruitment and dropout rates. Where possible, reasons for declining participation in the study and reasons for dropout will be documented. The ability of the patients to perform study related assessments will be recorded in addition to the reason for them being unable to perform the task, this will be done via a questionnaire that patients will complete at the end of each 3D biomechanical assessment session.

Patients will be asked to attend a biomechanical testing session before their surgery. After surgery they will follow standard aftercare, and on the day of discharge from the inpatient physiotherapy team they will be asked to attend the second biomechanical testing session. The third and fourth sessions will be on day three and day seven post-surgery, and the final session will take place when they return to the hospital for their standard three month follow up with the arthroplasty team. At the end of the three month visit, their involvement in the study will be complete.

Biomechanical movement analysis will be carried out in an on-site movement analysis laboratory. Study participants will be required to wear suitable clothing (e.g. tee shirt and shorts) and be barefoot. A number of reflective markers and surface electrodes will be attached to specific locations on the body using suitable double sided tape which can be tracked by a number of infrared cameras. participants will be asked to perform the following tasks; walking, sit-to-stand and stand-to-sit. Each task will be performed at least three times to enable the collection of three good sets of data. A motion capture system will collect limb and torso movements during the task performances while force plates will collect ground reaction forces.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for posterolateral approach total hip arthroplasty
* Able to give informed consentAble to return to study site for follow-up
* BMI under 35

Exclusion Criteria:

* Previous hip procedure in the previous twelve months
* Previous knee surgery other than arthroscopy and medial menisectomy in the last twelve months
* Symptomatic foot, knee, contralateral hip or spinal pathology
* Any medical condition limiting normal ambulation e.g. stroke, Parkinsons disease, severe lymphedema, advanced cardiac disease
* Unable to read and understand English and follow verbal and visual instructions unless they can bring a relative or friend to all study assessments to act as a translator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred to the Golden Jubilee National Hospital for total hip replacement.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Patient adherence to study procedures | 3 months
  Patients ability to attend for follow up appointments and carry out study specific biomechanical assessments

SECONDARY OUTCOMES:
Eligible patients | 1 year
  Number of suitable patients per consultant per month
Recruitment rate | 1 year
  Percentage of eligible patients recruited
Loss to follow up | 3 months
  Number of patients who choose to withdraw/ are lost to follow up
Hip angles during walking | 3 months
  Hip angles of movement collected using clinical movement analysis
Hip loads during walking | 3 months
  Hip loading collected using clinical movement analysis
Hip angles during sit to stand to sit | 3 months
  Hip angles of movement collected using clinical movement analysis
Hip loads during sit to stand to sit | 3 months
  Hip loading collected using clinical movement analysis
Muscle activation patterns walking | 3 months
  Hip muscle activation during level walking
Muscle activation patterns stand to sit to stand | 3 months
  Hip muscle activation during stand to sit to stand

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Ohly, MBBS, FRCSEd, Principal Investigator — Golden Jubilee National Hospital
Locations (1):
- Golden Jubilee National Hospital, Clydebank, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pabinger C, Lothaller H, Portner N, Geissler A. Projections of hip arthroplasty in OECD countries up to 2050. Hip Int. 2018 Sep;28(5):498-506. doi: 10.1177/1120700018757940. Epub 2018 May 21. PMID 29783896
- [Background] Lubbeke A, Katz JN, Perneger TV, Hoffmeyer P. Primary and revision hip arthroplasty: 5-year outcomes and influence of age and comorbidity. J Rheumatol. 2007 Feb;34(2):394-400. Epub 2006 Nov 15. PMID 17143967
- [Background] Hossain M, Parfitt DJ, Beard DJ, Darrah C, Nolan J, Murray DW, Andrew G. Does pre-operative psychological distress affect patient satisfaction after primary total hip arthroplasty? BMC Musculoskelet Disord. 2011 Jun 1;12:122. doi: 10.1186/1471-2474-12-122. PMID 21631923
- [Background] Mariconda M, Galasso O, Costa GG, Recano P, Cerbasi S. Quality of life and functionality after total hip arthroplasty: a long-term follow-up study. BMC Musculoskelet Disord. 2011 Oct 6;12:222. doi: 10.1186/1471-2474-12-222. PMID 21978244
- [Background] Nilsdotter AK, Isaksson F. Patient relevant outcome 7 years after total hip replacement for OA - a prospective study. BMC Musculoskelet Disord. 2010 Mar 11;11:47. doi: 10.1186/1471-2474-11-47. PMID 20222962
- [Background] Mayr E, Nogler M, Benedetti MG, Kessler O, Reinthaler A, Krismer M, Leardini A. A prospective randomized assessment of earlier functional recovery in THA patients treated by minimally invasive direct anterior approach: a gait analysis study. Clin Biomech (Bristol). 2009 Dec;24(10):812-8. doi: 10.1016/j.clinbiomech.2009.07.010. Epub 2009 Aug 21. PMID 19699566
- [Background] Stief F, Schmidt A, van Drongelen S, Lenarz K, Froemel D, Tarhan T, Lutz F, Meurer A. Abnormal loading of the hip and knee joints in unilateral hip osteoarthritis persists two years after total hip replacement. J Orthop Res. 2018 Mar 14. doi: 10.1002/jor.23886. Online ahead of print. PMID 29536559
- [Background] Bahl JS, Nelson MJ, Taylor M, Solomon LB, Arnold JB, Thewlis D. Biomechanical changes and recovery of gait function after total hip arthroplasty for osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2018 Jul;26(7):847-863. doi: 10.1016/j.joca.2018.02.897. Epub 2018 Feb 21. PMID 29474993
- [Background] Kolk S, Minten MJ, van Bon GE, Rijnen WH, Geurts AC, Verdonschot N, Weerdesteyn V. Gait and gait-related activities of daily living after total hip arthroplasty: a systematic review. Clin Biomech (Bristol). 2014 Jun;29(6):705-18. doi: 10.1016/j.clinbiomech.2014.05.008. Epub 2014 Jun 2. PMID 24951319
- [Background] Bennett D, Ryan P, O'Brien S, Beverland DE. Gait kinetics of total hip replacement patients-A large scale, long-term follow-up study. Gait Posture. 2017 Mar;53:173-178. doi: 10.1016/j.gaitpost.2017.01.014. Epub 2017 Jan 21. PMID 28171843
- [Background] Agostini V, Ganio D, Facchin K, Cane L, Moreira Carneiro S, Knaflitz M. Gait parameters and muscle activation patterns at 3, 6 and 12 months after total hip arthroplasty. J Arthroplasty. 2014 Jun;29(6):1265-72. doi: 10.1016/j.arth.2013.12.018. Epub 2013 Dec 18. PMID 24439753
- [Background] Longworth JA, Chlosta S, Foucher KC. Inter-joint coordination of kinematics and kinetics before and after total hip arthroplasty compared to asymptomatic subjects. J Biomech. 2018 Apr 27;72:180-186. doi: 10.1016/j.jbiomech.2018.03.015. Epub 2018 Mar 16. PMID 29576311
- [Background] Beaulieu ML, Lamontagne M, Beaule PE. Lower limb biomechanics during gait do not return to normal following total hip arthroplasty. Gait Posture. 2010 Jun;32(2):269-73. doi: 10.1016/j.gaitpost.2010.05.007. Epub 2010 Jun 11. PMID 20541940
- [Background] Lamontagne M, Beaulieu ML, Varin D, Beaule PE. Lower-limb joint mechanics after total hip arthroplasty during sitting and standing tasks. J Orthop Res. 2012 Oct;30(10):1611-7. doi: 10.1002/jor.22127. Epub 2012 Apr 16. PMID 22508467
- [Background] Palan J, Manktelow A. Surgical approaches for primary total hip replacement. Orthopaedics and Trauma. 2018;32(1):1-12.
- [Background] Dorr LD, Maheshwari AV, Long WT, Wan Z, Sirianni LE. Early pain relief and function after posterior minimally invasive and conventional total hip arthroplasty. A prospective, randomized, blinded study. J Bone Joint Surg Am. 2007 Jun;89(6):1153-60. doi: 10.2106/JBJS.F.00940. PMID 17545416
- [Background] Ewen AM, Stewart S, St Clair Gibson A, Kashyap SN, Caplan N. Post-operative gait analysis in total hip replacement patients-a review of current literature and meta-analysis. Gait Posture. 2012 May;36(1):1-6. doi: 10.1016/j.gaitpost.2011.12.024. Epub 2012 Mar 10. PMID 22410129
- [Background] Bernard J, Razanabola F, Beldame J, Van Driessche S, Brunel H, Poirier T, Matsoukis J, Billuart F. Electromyographic study of hip muscles involved in total hip arthroplasty: Surprising results using the direct anterior minimally invasive approach. Orthop Traumatol Surg Res. 2018 Dec;104(8):1137-1142. doi: 10.1016/j.otsr.2018.03.013. Epub 2018 May 16. PMID 29753876
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445